CLINICAL TRIAL: NCT04486911
Title: Pyrotinib Maleate, CDK4/6 Inhibitor and Letrozole in Combination for Treatment of Stage II-III Triple-positive Breast Cancer: a Phase II Clinical Trial
Brief Title: Pyrotinib Maleate, CDK4/6 Inhibitor and Letrozole in Combination for Stage II-III TPBC: a Phase II Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Professor, Shengjing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUKDEN01
Record Dates: First submitted 2020-07-21; First posted 2020-07-27 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; pyrotinib maleate; letrozole; CDK4/6 inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Combined Modality Therapy

STUDY DESIGN:
Intervention Model Description: single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib maleate, SHR6390, letrozole (Experimental): After providing written informed consent, the participants will undergo combined treatment of pyrotinib maleate, CDK4/6 inhibitor SHR6390, and letrozole. The effectiveness of the combined treatment will be evaluated by MRI every two treatment cycles. If the disease progresses, the participant will withdraw from the trial. If the combined treatment has identified effectiveness, the participant will undergo surgical treatment within 4 weeks (over 2 weeks) after termination of the neoadjuvant treatment. The patients will be followed up for 5 years.
  Interventions: Drug: Pyrotinib maleate, SHR6390, letrozole

INTERVENTIONS:
Drug: Pyrotinib maleate, SHR6390, letrozole — After providing written informed consent, the participants will undergo combined treatment of pyrotinib maleate, CDK4/6 inhibitor SHR6390, and letrozole. The effectiveness of the combined treatment will be evaluated by MRI every two treatment cycles. If the disease progresses, the participant will withdraw from the trial. If the combined treatment has identified effectiveness, the participant will undergo surgical treatment within 4 weeks (over 2 weeks) after termination of the neoadjuvant treatment. The patients will be followed up for 5 years.
  Other Names: combined treatment

SUMMARY:
The emergence of CDK4/6 inhibitors has brought hope to breast cancer patients resistant to endocrine therapy. In the mouse model, pyrotinib maleate combined with CDK4/6 inhibitor exhibits higher anti-tumor activity than any anti-tumor drug alone. Moreover, the toxicity of the combined therapy does not increase compared with monotherapy. This provides a good preclinical model for the treatment of breast cancer by pyrotinib maleate combined with CDK4/6 inhibitor. Based on above, it is hypothesized that pyrotinib maleate, CDK4/6 inhibitor SHR6390 and aromatase inhibitor letrozole in combination can provide a better neoadjuvant strategy for stage II-III triple-positive breast cancer.

DETAILED DESCRIPTION:
This single-center, single-arm, open-label trial will include 89 patients with stage II-III triple-positive breast cancer (Simon's two-stage design). After providing written informed consent, the participants will undergo combined treatment of pyrotinib maleate, CDK4/6 inhibitor SHR6390, and letrozole. The effectiveness of the combined treatment will be evaluated by MRI every two treatment cycles. If the disease progresses, the participant will withdraw from the trial. If the combined treatment has identified effectiveness, the participant will undergo surgical treatment within 4 weeks (over 2 weeks) after termination of the neoadjuvant treatment. The patients will be followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* (1)Women aged > 18 years and ≤ 80 years meeting one of the following conditions;

  1. Those previously receiving ovariectomy, or aged ≥ 60 years
  2. Those aged < 60 years who have had 12 consecutive months of amenorrhoea without any pathological or physical causes, and have postmenopausal E2 and follicle stimulating hormone (FSH) levels
  3. Premenopausal or perimenopausal women who are willing to receive LHRH agonist treatment during the study period
* (2) Women who have breast cancer histopathologically confirmed by positive estrogen receptor (ER; ≥ 10%), positive progesterone receptor (PR; ≥ 1%), and positive human epidermal growth factor receptor 2 (HER2) according to the 2018 American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) human epidermal growth factor receptor 2 (HER2) guideline. ER, PR and HER2 will be assessed by immunohistochemistry (IHC) on harvested tissue. ER, PR and HER2 will be considered positive if the IHC result is positive (score 3+), or the IHC result is positive (2+) and in situ hybridization (ISH) amplification rate (≥ 2.0);
* (3) Women having stage II-III breast cancer diagnosed based on AJCC cancer staging system (8th edition) who will be admitted because of breast cancer for the first time;
* (4) Karnofsky Performance Status (KPS) Scale score ≥ 70;
* (5) The functional level of organs must meet the following requirements:

  a) Bone marrow function i) Absolute neutrophil count ≥ 1.5 × 109/L (no use of growth factor within 14 days) ii) Platelet count ≥ 100 × 109/L (no corrective treatment within 7 days) iii) Hemoglobin level ≥ 100 g/L (no corrective treatment within 7 days) b) Liver and kidney function i) Total bilirubin ≤1 upper limit of normal value (ULN) ii) Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 3 × ULN (ALT and AST ≤ 5 × ULN in patients with liver metastasis) iii) Blood urea nitrogen (BUN) and creatinine ≤ 1.5 × ULN and creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula); c) Color Doppler echocardiography: Left ventricular ejection fraction ≥ 50% d) 12-lead electrocardiography: QTc interval ≤ 480 ms
* (6) Women who can undergo a biopsy;
* (7) Volunteers to participate in the study, provision of signed informed consent, good compliance and willingness to cooperate with follow-ups

Exclusion Criteria:

* (1) Women who have received any form of anti-tumor treatment - (chemotherapy, radiotherapy, molecular targeted therapy, or endocrine therapy);
* (2) Those who have received other anti-tumor drug treatments concurrently;
* (3) Those who have bilateral breast cancer, inflammatory breast cancer or occult breast cancer;
* (4) Those who have stage IV breast cancer;
* (5) Those who have breast cancer not histopathologically confirmed;
* (6) Those who have other malignant tumors (with the exception of healed cervical carcinoma in situ) occurring in the past 5 years;
* (7) Those who have severe dysfunction of the heart, liver, kidney, and other major organs;
* (8) There are multiple factors that affect drug administration and absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
* (9) Those who have participated in other clinical drug trials in the past 4 weeks;
* (10) Those who are known to have a history of allergy to the component of study drugs; those who have a history of immunodeficiency, including positive detection of human immunodeficiency virus, hepatitis C virus, active hepatitis B or other acquired, congenital immunodeficiency diseases, or organ transplantation;
* (11) Those who had suffered from any heart disease, including arrhythmia which requires drug treatment or is of clinical significance; myocardial infarction; heart failure; and any other heart disease judged by the investigator as unsuitable for this trial;
* (12) Pregnant and lactating women; fertile women who provide positive results of baseline pregnancy test; women of childbearing age who are unwilling to take effective contraceptive measures during the whole study period;
* (13) If the accompanying diseases (including, but not limited to, severe hypertension, severe diabetes, and active infection, which cannot be controlled by drugs) that would be a potential hazard to participant's health, or affect the completion of the study as per investigator's judgement;
* (14) A clear history of neurological or psychiatric disorders, including epilepsy or dementia;
* (15) Upon the suggestion of the investigators for other reasons

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Total pathological complete response (tpCR) | 1 month to 5 years after surgery
  tpCR is defined as the absence of residual invasive cancer on resected breast specimen and the sampled regional lymph nodes as shown by hematoxylin-eosin staining after completion of the neoadjuvant treatment.

SECONDARY OUTCOMES:
Best overall response rate (BORR) | During neoadjuvant treatment (1-5 months of treatment)
  The proportion of patients who respond to the treatment at any study time point
Residual cancer burden (RCB) | 1 month to 5 years after surgery
  RCB score is obtained according to pathological evaluation after completion of neoadjuvant treatment and surgery
Change From Baseline of Functional Scales, Symptom Scales and Single Items in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Core 30 (QLQ-C30) | Baseline, the end of cycle 2, cycle 4, and before the surgery
  The EORTC QLQ-C30 included global health status, functional scales (physical, role, emotional, cognitive, and social), symptom scales (fatigue, nausea/vomiting, and pain) and single items (dyspnoea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Most questions used a 4-point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale [1 'very poor' to 7 'Excellent']). Scores were averaged and transformed to 0 - 100 scale, whereby higher scores indicate greater functioning, greater quality of life, or a greater degree of symptoms, with changes of 5 - 10 points considered to be a minimally important difference to participants. A positive value means an increase, while a negative value means a decrease, in score at the indicated time-point(the end of cycle 2, cycle 4, and before the surgery) relative to the score at baseline .
Change From Baseline of Four Functioning Scales and Four Symptom Scales in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Breast Cancer (QLQ-BR23) | Baseline, the end of cycle 2, cycle 4, and before the surgery
  EORTC-QLQ-BR23 is a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30 and consists of four functional scales (body image, sexual enjoyment, sexual functioning, future perspective [FP]) and four symptom scales (systemic side effects [SE], upset by hair loss, arm symptoms, breast symptoms). Questions used 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Scores averaged and transformed to 0-100 scale. High score for functional scale indicated high/better level of functioning/healthy functioning. Higher scores for symptom scales represent higher levels of symptoms/problems. For functional scales, positive change from baseline indicated deterioration in quality of life (QOL) and negative change from baseline indicated an improvement in QOL. For symptom scales, positive change from baseline indicated an improvement in quality of life (QOL) and negative change from baseline indicated a deterioration in QOL.

OTHER OUTCOMES:
Overall survival (OS) | Within 5 years after surgery
  It refers to the length of time from the start of treatment to the death of the patient.
Disease-free survival (DFS) | Within 5 years after surgery
  It refers to the length of time from the start of medication after enrollment to the death of the patient because of the recurrence, distant metastasis of the disease, invasive contralateral breast cancer, or any other cause.

CONTACTS AND LOCATIONS:
Overall Officials: Cai-Gang Liu, MD, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
Findings from this study will indicate whether pyrotinib maleate, CDK4/6 inhibitor SHR6390 and letrozole for treatment of stage II-III triple-positive breast cancer is safe and effective.
Supporting Information: Study Protocol
Time Frame: 6 months to 5 years after publication
Access Criteria: Unlimited

REFERENCES:
- [Derived] Bu J, Zhang Y, Niu N, Bi K, Sun L, Qiao X, Wang Y, Zhang Y, Jiang X, Wang D, Ma Q, Li H, Liu C. Dalpiciclib partially abrogates ER signaling activation induced by pyrotinib in HER2+HR+ breast cancer. Elife. 2023 Jan 5;12:e85246. doi: 10.7554/eLife.85246. PMID 36602226